CLINICAL TRIAL: NCT06258200
Title: Examining the Role of Gender Transformative Community Interventions to Strengthen Gender Equity and Improve Immunization Outcomes in Togo and Pakistan
Brief Title: The Role of Gender Transformative Interventions to Strengthen Gender Equity and Improve Immunization Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Gavi, The Vaccine Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00027395
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Gender Equality and Its Impact on Immunization Uptake
MeSH Terms: interventions — Sex

STUDY DESIGN:
Intervention Model Description: The study will have two arms, an intervention and comparison arm, and participants will be grouped into arms based on their community of residence. Participants in the intervention arm will receive behavioral interventions, including household visits, participation in couple discussion groups, and messaging from community leaders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this arm will receive behavioral interventions, including household visits, participation in couples discussion groups, and messaging from community leaders.
  Interventions: Behavioral: Gender and immunization activities
- Comparison (Experimental): Participants in this arm will not receive any interventions.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Gender and immunization activities — Household visits from community mobilizers, participation in couples communication groups, and messaging from community leaders.
  Arms: Intervention group
Other: No intervention — Participants in the comparison group will not receive any intervention
  Arms: Comparison

SUMMARY:
The goal of this clinical trial is to test the role of community-based men's engagement interventions in improving immunization uptake and strengthening gender equity at the household level. The main questions it aims to answer are: (1) Does household and community engagement of male caregivers and couples improve equitable gender relations, including increased male involvement in household tasks and childcare, in Togo and Pakistan, compared with communities that did not receive an intervention? (2) Can household and community engagement of male caregivers and couples increase support for and rates of age-appropriate timely immunization among children under 12 months of age, in Togo and Pakistan, compared with communities that did not receive an intervention? (3) How feasible, acceptable, and appropriate is it for CSO staff/volunteers to engage female and male caregivers and community leaders using gender transformative approaches (including household visits and group discussions) as assessed over a seven-month period? (4) What is the cost of gender transformative engagement of male and female caregivers and community leaders by CSO staff/volunteers compared to standard childhood immunization outreach services over a seven-month period?

Participants (male and female caregivers of children under 12 months of age) will be sorted into intervention or comparison groups based on their community of residence. Participants in the intervention group will:

* Receive household visits to raise awareness of immunization benefits and gender equity
* Participate in couples communication discussion groups
* Receive immunization and gender equity messaging from community leaders and other influencers.

Researchers will compare the intervention group with comparison groups in similar communities to see if the intervention group demonstrates improved equitable gender relations and increased rates of immunization compared to the comparison group which does not receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

Caregivers Pakistan:

* Adult women and men aged 18-49 who are in a monogamous relationship, or polygamous relationship in which the male partner agrees to participate with one female partner, and are together caregivers of at least one child 12 months of age or younger
* Have lived in the study site for at least one year
* Plan to continue to live in the study site for at least one year from time of recruitment
* If the caregiver is drawn from one of the intervention Union Councils, must be willing to fully participated in the intervention for the full implementation period

Caregivers Togo:

* Adult women and men aged 18-49 who are in a monogamous relationship, or are in a polygamous relationship in which the man resides only with the woman who is also involved in the study, and who and are together caregivers of at least one child 12 months of age or younger
* Have lived in the study site for at least one year
* Plan to continue to live in the study site for at least one year from time of recruitment
* If the caregiver is drawn from one of the intervention communities, must be willing to fully participate in the intervention for the full implementation period

Community mobilizers Pakistan:

* A woman or man currently living in the intervention Union Councils
* Has at least one child who has received the complete vaccine series
* Fluently speak the language that is most commonly spoken in the Union Council in which they live
* Be able to read and write
* Have previous experience of working on advocacy and community mobilization
* Have previously worked on childhood immunization mobilization
* Are familiar with the community influencers
* Are willing to complete training for the intervention
* Must be willing to actively implement intervention for the full implementation period

Papas Champions Togo:

* Be a married man with children, who has demonstrated his involvement in his children's health
* Has at least one child who has received the complete vaccine series
* Currently live in the intervention community
* Fluently speak the language that is most commonly spoken in the community in which they live
* Be able to read and write
* Be willing to promote the benefits of vaccination to other fathers in the community
* Be willing to work on a voluntary basis*
* Be accepted by the local community and recognized as a responsible and respectable person.
* Be willing to complete training for the intervention
* Be willing to actively implement the intervention for the full implementation period

CSO Leaders Pakistan:

* Be based in one of the intervention Union Councils
* Actively support implementation intervention

CSO Leaders Togo:

* Be based in one of the intervention districts
* Actively support implementation intervention

Community Leaders Pakistan:

* Be based in one of the intervention Union Councils
* Have known influence on gender dynamics, caregiving, and child health behaviors including immunization
* Be willing to participate in the values clarification and attitudinal transformation activities conducted as part of the intervention

Community Leaders Togo:

* Be based in one of the intervention communities
* Have known influence on gender dynamics, caregiving, and child health behaviors including immunization
* Be willing to participate in the community sensitization activities conducted as part of the intervention

EPI Stakeholders Pakistan/Togo:

* Be based in one of the study districts since the beginning of the study
* Be familiar with the operations research intervention conducted as part of the study

Exclusion Criteria:

Any individuals that do not meet all of the above inclusion criteria or do not agree to participate in the study will be excluded from data collection. In addition, individuals who are unable to make decisions/respond to questions on their own without assistance by someone else will also be excluded from enrolment.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 448 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sharing of childcare and household tasks | 7 months
  Administered to all male caregivers via survey, sample of female caregivers via FGDs:
  How do you divide the following childcare and household tasks: (1) washing clothes/laundry; (2) cleaning the house and surroundings; (3) cooking for the household; (4) making the bed; (5) providing daily care of children; (6) bathing children. [Gendered division of household labor]
  Responses range from 1 = woman always does the task, 3 = shared equally or done together, 5 = man always does the task.

SECONDARY OUTCOMES:
Couples' communication | 7 months
  Administered to all male caregivers via survey, sample of female caregivers via FGDs:
  In the last three months, how many times have you discussed with your partner about immunizing your child, and offered your opinion about immunizing your child as part of the discussion? [MOMENTUM]
  Responses range from 0 = never, 1 = rarely (1-2 times), 2 = sometimes (3-5 times), 3 = a lot (6 or more times)
Decision-making about child health practices, including vaccination | 7 months
  Administered to all male caregivers via survey, sample of female caregivers via FGDs:
  Did you take part in the decision to immunize your child? [Adapted from Galle et al, 2011]
  Responses range from 1 =I was the sole decision-maker; 2 = I made the decision jointly with my partner; 3 = I made the decision jointly with someone else; 4 = My partner was the sole decision-maker
Vaccination uptake | 7 months
  Review of vaccine cards or interviewee responses for date of the following vaccines:
  * Penta 1 (six weeks)
  * Penta 3 (14 weeks)
  * MCV 1 (9 months)
  * MCV 2 (15 months)
Acceptability of intervention | Pre/post test: prior to intervention, as part of implementer training (month zero); pulse surveys: monthly; Lessons learned workshop: Month 4
  Measured through monthly pulse surveys to community mobilizers, through pre/post tests during the training of community mobilizers, and through a lessons learned workshop at the end of the intervention.
Appropriateness of the intervention | Pulse surveys: monthly; Lessons learned workshop: Month 4
  Measured through monthly pulse surveys administered to community mobilizers as well as a lessons learned workshop immediately following the intervention
Feasibility of the intervention | Pre/post test: prior to intervention, as part of implementer training (month zero); pulse surveys and supervision data: monthly; Lessons learned workshop: Month 4
  Measured through monthly pulse surveys to community mobilizers, through pre/post tests during the training of community mobilizers, monthly supervision data, and through a lessons learned workshop at the end of the intervention
Cost of intervention | Months 1-4
  This will include analysis of:
  * CSO costs
  * Technology support costs
  * Materials and training costs
  * Other costs as appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Charurat, Study Director — Jhpiego
Locations (19):
- Pakistan (4):
  - Community Setting, Uc-10 Pehalwan Goth - Gulshan Town, Karachi East
  - Community Setting, Uc-11 Garden East - Jamshed Town, Karachi East
  - Community Setting, UC 10/B, Quetta
  - Community Setting, UC 13/A, Quetta
- Togo (15):
  - Community Setting, Adakpamé, Golfe
  - Community Setting, Adamavo, Golfe
  - Community Setting, Kanyikope, Golfe
  - Community Setting, Ségbé, Golfe
  - Community Setting, Gbodjome / Kpogan Agbetiko, Lacs
  - Community Setting, Gbodjome /agbataloglo, Lacs
  - Community Setting, Moretan /assati, Mono-Est
  - Community Setting, Kpekpleme/ Kativou, Moyen-mono
  - Community Setting, TADO /tado DOME, Moyen-mono
  - Community Setting, Dagbati, Vo
  - Community Setting, Dzrekpo /klologo, Vo
  - Community Setting, Ahépé, Yoto
  - Community Setting, Kouvé, Yoto
  - Community Setting, Abobo / LEBE, Zio
  - Community Setting, Mission TOVE / Apessito, Zio

IPD SHARING:
Plan to Share IPD: No
The de-identified data set will be uploaded in an online repository accessible to other researchers.